CLINICAL TRIAL: NCT01654068
Title: Conformal High Dose Intensity Modulated Radiation Therapy for Asymptomatic Metastatic Disease to the Thoracic and Lumbar Spine
Brief Title: Conformal High Dose Intensity Modulated Radiation Therapy for Disease to Thoracic and Lumbar Spine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low participant accrual
Sponsor: Ronald McGarry (Other)
Responsible Party: Sponsor-Investigator, Ronald McGarry, Professor, Radiation Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-09-RAD-01
Record Dates: First submitted 2012-07-17; First posted 2012-07-31 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-03

CONDITIONS: Vertebral Metastasis
Keywords: Female Breast Cancer; Kidney Cancer; Lung Cancer; Prostate Cancer; Vertebral metastasis
MeSH Terms: conditions — Kidney Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Molecular Conformation; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation Therapy to Local Spine Metastasis (Experimental): Conformal High Dose Intensity Modulated Radiation Therapy to a single asymptomatic local spine metastasis.
  Interventions: Radiation: Conformal High Dose Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Conformal High Dose Intensity Modulated Radiation Therapy — Conformal High Dose Intensity Modulated Radiation Therapy 14-16Gy single fraction dosing using 6MV photons

SUMMARY:
The purpose of this study is to determine if Conformal High Dose Intensity Modulated Radiation Therapy is an appropriate option for treating cancer that has spread to the spinal column. This study involves patients who have been diagnosed with metastatic cancer to the thoracic and lumbar vertebral body levels and currently do not have symptoms caused from the area of concern. The goal is to prove that this is not only a safe form of treatment, but that Conformal High Dose Intensity Modulated Radiation Therapy can reduce the risk of cancer coming back in the area that the investigators treat which may reduce the risk of developing symptoms like pain in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of malignancy (non-small cell lung cancer, breast cancer (hormone refractory), prostate cancer (hormone refractory), lymphoma, renal cell carcinoma, myeloma by either biopsy or cytology of the primary or metastatic lesion.
* Patients must have radiological documentation of metastatic disease to the thoracic or lumbar spine including both positron emitted tomography (PET) or nuclear medicine bone scan (NMBS) and Magnetic Resonance Imaging (MRI) within 4 weeks prior to study entry.
* Patients with one to three spinal metastases to the thoracic or lumbar spine will be included.
* Spinal metastatic lesions should be limited to one vertebral body level or ≤ 6cm in greatest dimension.
* Tumors should not directly abut the spinal cord, and have at least 5mm separation from the spinal cord. For patients with tumors closer than 5mm, inclusion is permissible at the discretion of the treating radiation oncologist such that dosimetric review demonstrates that the total dose to spinal cord is within tolerable range of <10Gy to 10% partial volume or max point dose 18 Gy.
* Patients must be able to fit into either the Elekta Stereotactic Body Frame or the Elekta Stereotactic BodyFix immobilization device.
* Must be ≥ 18 years of age.
* ECOG status 0-2.
* Women of childbearing potential and male participants must use an effective contraception method. (Until at least 60 days following treatment.)
* Negative urine pregnancy test within at least one week before starting treatment in women of child-bearing age.
* Patients must sign a study-specific informed consent form.

Exclusion Criteria:

* Patients with evidence of spinal instability OR neurologic deficit resulting from bony compression of neurologic structures.
* Patients with other systemic illness, or have not recovered adequately from their primary treatment or who have evidence of progression of their current cancer prior to therapy that, in the investigator's opinion, would preclude their inclusion.
* Patient may not receive concomitant cytotoxic anti-neoplastic therapy during treatment. Patients may be allowed to use hormonal suppression therapy or bisphosphonates for hypercalcemia.
* Pregnant or lactating women.
* Any patient with symptoms of pain, compression fracture, neurologic deficit will not be included.
* Patients previously treated with radiation therapy to the thoracic or lumbar spinal levels of involved disease will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald McGarry, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy to Local Spine Metastasis: Conformal High Dose Intensity Modulated Radiation Therapy
  Conformal High Dose Intensity Modulated Radiation Therapy: Conformal High Dose Intensity Modulated Radiation Therapy 14-16Gy single fraction dosing using 6MV photons
Period: Overall Study
Arm/Group | Radiation Therapy to Local Spine Metastasis
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy to Local Spine Metastasis
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 66 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 14
Smoking Status [Count of Participants; unit: Participants]
  Never Smoker | 5
  Former Smoker | 8
  Current Smoker | 1
Site of Metastasis [Count of Participants; unit: Participants]
  Thoracic Spine | 10
  Lumbar Spine | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Any Skeletal Related Event
Description: Time to any skeletal related event most commonly symptomatic recurrence or progression with pain/neurologic impairment with evidence of radiographic progression (median local progression-free survival).
Time Frame: up to 24 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Radiation Therapy to Local Spine Metastasis
Number analyzed (Participants) | 14
weeks | 75 [33 to 75]

2. Secondary Outcome: Acute Radiation Toxicity
Description: The number of acute side effects of radiation therapy will be documented (≤ 90 days from start of radiation therapy)
Time Frame: 90 days
Measure: Number; unit: event (possible acute side effect)
Arm/Group | Radiation Therapy to Local Spine Metastasis
Number analyzed (Participants) | 14
event (possible acute side effect) | 1

3. Secondary Outcome: Late Radiation Toxicity
Description: The number of late side effects of radiation therapy will be documented (> 90 days after the start of radiation therapy)
Time Frame: 2 years
Measure: Number; unit: events (possible late side effects)
Arm/Group | Radiation Therapy to Local Spine Metastasis
Number analyzed (Participants) | 14
events (possible late side effects) | 2

ADVERSE EVENTS:
Time Frame: 0-209 weeks
Arm/Group | Radiation Therapy to Local Spine Metastasis
All-Cause Mortality (participants affected / at risk) | 11/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy to Local Spine Metastasis (N=14)
Vertebral Compression Fractures (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy to Local Spine Metastasis (N=14)
Bilateral Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-06-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT01654068/Prot_SAP_000.pdf
  • Informed Consent Form (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT01654068/ICF_001.pdf